CLINICAL TRIAL: NCT02334397
Title: Bump on the Ball: Impact of a Prenatal Exercise & Education Program on Birth Outcomes & Maternal Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Christina Lewicky-Gaupp, Assistant Professor of Obstetrics and Gynecology, Associate Residency Program Director, Medical Director of PEAPOD clinic, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STU00095770
Record Dates: First submitted 2015-01-05; First posted 2015-01-08 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy
Keywords: Prenatal Exercise; Prenatal Education; Pregnancy; Exercise and Birth Outcomes; Education and Birth Outcomes; Maternal Quality of Life; Birth Satisfaction
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Control Program (Active Comparator): Women will be enrolled in Total Control, which is a fitness and education program. Specifically, Total Control is a comprehensive pelvic fitness and wellness program designed by board-certified female pelvic medicine and reconstructive surgery (FPMRS) practitioners as well as physical therapists that combines pelvic floor and core muscle strengthening. Subjects will participate in 1 standardized class per week during their second trimester for a total of 6 weeks. Women will also participate in a weekly educational session which will include keynote speakers who are experts in various aspects of the labor and delivery process. Women in this group will complete questionnaires and consent to use of their delivery outcomes. Women will also wear pedometers to track daily general activity.
  Interventions: Behavioral: Total Control Program
- Control Group (No Intervention): This group will consist of eligible women who were not randomized to the fitness and education program. Participants will complete questionnaires and consent to use of their delivery outcomes. Women will also wear pedometers to track daily general activity.

INTERVENTIONS:
Behavioral: Total Control Program — Women will be enrolled in Total Control, which is a fitness and education program.
  Arms: Total Control Program

SUMMARY:
Operative vaginal delivery (with forceps or vacuums) is frequently performed secondary to maternal exhaustion, which leads to an inability to push effectively; 40% of operative vaginal deliveries at Prentice are for maternal exhaustion. The risk of severe birth trauma is increased three to four fold with operative delivery. This randomized, controlled trial will compare rates of operative vaginal delivery and severe birth trauma in two groups of women: (1) an intervention group who will participate in the antepartum Total Control® fitness and education program modified for pregnancy; and (2) a control group. Women will be recruited and followed from the second trimester until 6 weeks postpartum; all will complete validated questionnaires regarding their (1) level of worry and knowledge about their birthing experience (2) pelvic floor symptoms and quality of life (3) sexual function (4) satisfaction with their birthing experience and (5) level of depressive symptoms at various time points during and after their pregnancy. Obstetrical data will also be collected.

DETAILED DESCRIPTION:
This will be a randomized controlled trial of primiparous women with singleton pregnancies who plan on delivering at Prentice Women's Hospital. Women will be recruited during their first trimester by their obstetrician as well as through standardized Northwestern Memorial Hospital flyers and ads. Demographic and delivery information will be obtained from the Northwestern Enterprise Data Warehouse (EDW), as well as by the attending midwife or physician at the time of delivery using a standardized Delivery Information Form. Women will also be asked about their other physical activities (including other forms of daily/weekly exercise) as well as whether or not they are participating in other birthing classes at the time of their first Total Control class (intervention group) or 2nd trimester visit with their providers (controls). All women will wear pedometers to track daily general activity.

ELIGIBILITY:
Inclusion Criteria:

* Singleton, primiparous pregnancy
* Delivering at Prentice Women's Hospital
* Able to participate based on PARmedX for pregnancy criteria

Exclusion Criteria:

* Non-english or Spanish speaking
* Age less than 18 years
* Known condition requiring cesarean section
* Currently enrolled in any kind of physical therapy
* Unable to complete the program secondary to medical limitations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02; Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Predomination of type of birth, operative vaginal delivery versus natural spontaneous vaginal delivery | At time of delivery (~6 months after baseline)
  We will be comparing the proportion of women who undergo operative vaginal delivery versus natural spontaneous vaginal delivery among pregnant women participating in an antepartum fitness and education program and women not participating in the program. We will do so using standard Delivery Information Forms and Northwestern University's Electronic Data Warehouse (EDW).
Indication for operative vaginal delivery (if applicable) | At time of delivery (~6 months after baseline)
  We will compare the indication for operative vaginal delivery among women who undergo operative vaginal deliveries. We will do so using standard Delivery Information Forms and Northwestern University's Electronic Data Warehouse (EDW).

SECONDARY OUTCOMES:
Obstetrical Complications (using data from Northwestern's Electronic Data Warehouse) | From time of delivery to 6 weeks Postpartum
  We will be comparing both groups' obstetrical complications, including rates of severe perineal trauma or obstetrical anal sphincter lacerations and wound complications, among intervention and control groups. We will do so using data from Northwestern's Electronic Data Warehouse (EDW).
Level of worry/concern about the birthing experience (Penn State Worry Questionnaire) | Baseline, at time of delivery, 6 weeks postpartum
  Penn State Worry Questionnaire (PSWQ) scores will be compared among the groups to determine which group will have less worry/concern about their birthing experience.
Knowledge about the birthing experience ( Birth Technology and Maternal Roles in Birth: Knowledge and Attitudes of Canadian Women Approaching Childbirth for the First Time Questionnaire) | Baseline, at time of delivery, 6 weeks postpartum
  Knowledge about the birthing experience will be compared between groups utilizing the Birth Technology and Maternal Roles in Birth: Knowledge and Attitudes of Canadian Women Approaching Childbirth for the First Time Questionnaire (KA)
Pelvic Floor Symptoms (Pelvic Floor Distress Inventory) | Baseline, at time of delivery, 6 weeks postpartum
  Baseline and postpartum pelvic floor symptoms will be compared between groups using the short form of the Pelvic Floor Distress Inventory (PFDI-SF).
Sexual Function (Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) | Baseline, at time of delivery, 6 weeks postpartum
  Baseline and postpartum sexual function will be compared between groups using the Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12)
Satisfaction with birthing experience (Satisfaction with Childbirth Rating Scale (SatCh) and Mackey Satisfaction with Childbirth Rating Scale) | At time of delivery and during 6 weeks postpartum
  Satisfaction with the birthing experience will be compared among intervention and non intervention groups utilizing the Satisfaction with Childbirth Rating Scale (SatCh) and Mackey Satisfaction with Childbirth Rating Scale
Postpartum Depression Incidence and Risk Factors ( Edinburgh Postnatal Depression Scale) | 6 weeks postpartum
  Incidence of and risk factors for postpartum depression will be compared between groups using the Edinburgh Postnatal Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Gaupp, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Medical Group's Integrated Pelvic Health Program, Chicago, Illinois, United States

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735